CLINICAL TRIAL: NCT05184972
Title: Coverage and Validity of the Swedish Registry of Cardiopulmonary Resuscitation Regarding In-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Dalarna University (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Jennie Silverplats, PhD student, Dalarna University
Other Study IDs: 2021-04102
Record Dates: First submitted 2021-12-08; First posted 2022-01-11 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: In-hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-reported patients treated for in-hospital cardiac arrest
- Reported patients treated for in-hospital cardiac arrest

SUMMARY:
The study will have an observational retrospective cross-sectional design. Patient records and hospital administrative systems at 10 hospitals in Sweden will be searched using ICD-codes to find all patients treated for an in-hospital cardiac arrest (IHCA) during the time period of 20180101 to 20191231. All found patients will be cross-checked against reported patients in the Swedish Registry of Cardiopulmonary Resuscitation (SRCR). Any differences in patient characteristics or regarding situation factors between reported and non-reported patients will be evaluated. Non-reported patients will be retrospectively reported to the registry. An incidence of IHCA will be calculated using the number of patients treated for IHCA divided by number of hospital admissions during the specific time period. Selected variables will be evaluated regarding compliance to report and regarding concordance with patient records. All missing data will be described and evaluated. Local reporting procedures at each hospital will be described and evaluated regarding compliance to report and regarding missing data.

ELIGIBILITY:
Inclusion Criteria:

* All patients after the neonatal period that have been treated for an in-hospital cardiac arrest.

Exclusion Criteria:

* Patients with an in-hospital cardiac arrest that is not treated (do not attempt resuscitation) or patients in the neonatal period.

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An in-hospital cardiac arrest is defined as an arrest that occurs in a hospitalized patient who had a pulse at the time of admission. A hospital is defined as a facility with twenty-four hours a day care including an intensive care unit and an emergency team. Treatment of a cardiac arrest involves initiation of CPR or defibrillation. Data of patients treated for in-hospital cardiac arrest will be collected from 10 hospitals of varying size during 20180101 to 20191231 in Sweden. Data of reported patients treated for in-hospital cardiac arrest during the same time period at each hospital will be extracted from the SRCR .
Sampling Method: Probability Sample
Enrollment: 1109 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Proportion of reported patients treated for in-hospital cardiac arrest | During hospital stay (retrospective observation january 1 2018 to december 31 2019)
  To evaluate the proportion of patients treated for in-hospital cardiac arrest that are reported to the SRCR

SECONDARY OUTCOMES:
Incidence of in-hospital cardiac arrest | During hospital stay (retrospective observation january 1 2018 to december 31 2019)
  To calculate an incidence of number of patients treated for in-hospital cardiac arrest based on number of hospital admissions during a specific time period.
Patient characteristics | During hospital stay (retrospective observation january 1 2018 to december 31 2019)
  To evaluate possible differences in patient characteristics or situation factors between reported and non-reported patients treated for in-hospital cardiac arrest.

OTHER OUTCOMES:
Reporting procedures at hospitals | At study start (interview with CPR coordinators)
  To describe reporting procedures at each hospital in relation to coverage of patients treated for in-hospital cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Strömsöe, PhD, Principal Investigator — Dalarna University
Locations (1):
- Registercentrum Västra Götaland, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No